CLINICAL TRIAL: NCT02671344
Title: Determination of Gene Profiling in Semen Donors With Pregnancy Versus no Donor Gestation, Obtained in Assisted Reproduction Treatments
Brief Title: Determining the Genetic Profile in Semen Donors With Pregnancy, Donor Versus no Pregnancy Obtained in TRA
Status: Terminated | Type: Observational
Why Stopped: could not be obtained enough sperm RNA is highly fragmented and very difficult to purify.
Sponsor: IVI Bilbao (Other)
Collaborators: Fundación IVI (Other)
Responsible Party: Sponsor
Other Study IDs: 1406-BIO-036-FQ
Record Dates: First submitted 2016-01-25; First posted 2016-02-02 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Donor Site Complication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Determination of gene profiles characterizing the set of mRNA from donor seminal samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- IAD group: Sperm donors from donation program who have obtained three pregnancies Sperm donors from donation program that have not generated gestation IAD group 'Determination of gene profiles using arrays semen'
  Interventions: Other: Determination of gene profiles using arrays semen
- FIV group: Sperm donors from donation program who have obtained three pregnancies Sperm donors from donation program that have not generated gestation FIV group of gene profiles using arrays semen'
  Interventions: Other: Determination of gene profiles using arrays semen
- ICSI group: Sperm donors from donation program who have obtained three pregnancies Sperm donors from donation program that have not generated gestation 'Determination of gene profiles using arrays semen'
  Interventions: Other: Determination of gene profiles using arrays semen

INTERVENTIONS:
Other: Determination of gene profiles using arrays semen — Determination of gene profiles characterizing the set of mRNA and functional interpretation of the resulting list of genes.

SUMMARY:
Microarray experiments to assess the expression of thousands of genes providing vast amount of information.

Because the molecular requirements in the different processes related to playback,on the hypothesis that there may be more apt semen samples for technical or other assuming molecular differences in RNA content messengers or gene expression profile between the They getting semen samples in gestation versus those who do not.

In an attempt to give a functional data obtained view, it is to find out how many of these genes in donors who have obtained gestation, they are differentially expressed in playback related processes against those donors who did not get pregnant.

DETAILED DESCRIPTION:
MRNA assembly is characterized by using microarrays on semen samples from donors included in the donation program of the clinic.

This process is performed in donors who have generated at least 3 pregnancies compared those samples, however, were not a function of gestation assisted reproduction technique used.

Consequently, differential expression of genes are identified in assisted reproduction treatment cycles from IAD, IVF or ICSI.

ELIGIBILITY:
Inclusion Criteria:

IAD group Younger than 37 years, natural cycles and stimulated apparently no problem of infertility as follows:

* Polycystic ovary syndrome.
* Endometriosis.
* ovarian failure.
* Lack of tubal patency (Both fallopian tubes must submit permeability).
* altered hormonal profiles (High levels of FSH, LH, testosterone and androstenedione).
* Anovulation.
* Uterine malformations (uterine septum, bicorne, didelphic and unicorn.)
* Ovarian cysts or tumors.
* Pelvic inflammatory disease.
* Obesity (Women with a BMI> 30).
* Thyroid Disease.
* Diabetes mellitus.
* renal or adrenal disease.
* toxic habits (smoking, alcohol or drug abuse).

IVF group Couples who undergo IVF egg donation invoking the program. Therefore, they try to cycles in which two gametes were donors. All egg donors should be fertility proven, it is that must have been able to take shape within the program of egg donation or naturally. The recipient women (patients) should not present

* Endometriosis.
* Uterine malformations (uterine septum, bicorne, didelphic and unicorn.)
* previous implantation failures.
* cysts, polyps or uterine tumors.
* Pelvic inflammatory disease.
* Obesity (Women with a BMI> 30)
* Thyroid Disease.
* Diabetes mellitus. Renal or adrenal disease,
* toxic habits (smoking, alcohol or drug abuse)

ICSI group Couples who undergo ICSI invoking the egg donation program. In addition, all donors oocytes must be of proven fertility, this being that should have been able to take shape within the egg donation program or naturally. The recipient women (patients) should not present

* Endometriosis.
* Uterine malformations (uterine septum, bicorne, didelphic and unicorn.)
* previous implantation failures.
* cysts, polyps or uterine tumors.
* Pelvic inflammatory disease.
* Obesity (Women with a BMI> 30)
* Thyroid Disease.
* Diabetes mellitus. Renal or adrenal disease,
* toxic habits (smoking, alcohol or drug abuse)

Exclusion Criteria:

-

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Open retrospective study of 30 semen donors. Comparisons were made of gene expression profile between the IAD, IVF and ICSI groups according to the clinical outcomes of pregnancy.
  * The donor recruitment will be made according to standard protocols rather Bilbao IVI centers will no visit, checking out additional analytical donation program to the donor is attached.
  * By SIVIS data base, the results of different gestation is collected reproductive treatments that allow the allocation to the comparison groups gene profile.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Detecting gene expression differences in RNA content messengers or gene expression profile between the semen samples versus those who get pregnant when you do not. | 15 months
  mRNA whole is characterized by using microarrays, in semen samples from donors included in the donation program of the clinic.
  By using bioinformatics tools Gene Ontology search listings of genes related to reproduction for the interpretation and identification of those who are involved in the different processes will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Quintana, Principal Investigator — IVI Bilbao
Locations (1):
- IVI Bilbao, Leioa, Vizcaya, Spain

IPD SHARING:
Plan to Share IPD: Undecided